CLINICAL TRIAL: NCT00888797
Title: Perioperative β-adrenergic Blocker and a COX2 Inhibitor in Patients Undergoing Resection for Primary Colon and Rectal Cancer: Effect on Tumor Recurrence and Postoperative Immune Perturbations. A Multicenter Randomized Prospective Trial.
Brief Title: β-adrenergic Blocker and a COX2 Inhibitor for Prevention of Colorectal Cancer Recurrence
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government); Rabin Medical Center (Other)
Responsible Party: Oded Zmora, MD, Deparetment of Surgery, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SHEBA-09-6994-OZ-CTIL
Record Dates: First submitted 2009-04-26; First posted 2009-04-28 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Propranolol; Etodolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Perioperative Propranolol and Etodolac
  Interventions: Drug: Propranolol and Etodolac
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Propranolol and Etodolac

INTERVENTIONS:
Drug: Propranolol and Etodolac — Both study medications will be given orally for an intervention phase of 20 days as follows: 5 days prior to surgery, on the day of surgery, and 14 days postoperatively. Etodolac:800 mg PO bid for the entire intervention period,Propranolol:20 mg PO bid for 5 preoperative days, 80 mg PO bid on the day of surgery, 40 mg PO bid for the first postoperative week, 20 mg PO bid for the second postoperative week.

SUMMARY:
Colon and rectal cancer is the second most prevalent malignant disease in the western world, causing significant morbidity, mortality, and healthcare sources use. Treating colon and rectal cancer with curative intent generally includes resection of the primary tumor. Despite its crucial role, surgery by itself induce physiological changes resulting in significant immune depression and other physiological perturbations, which may in turn play a significant role in the initiation of new metastases and the progression of pre-existing dormant metastases. The aim of this study is to assess the use of perioperative medical intervention using a combination of a β-adrenergic blocker (Propranolol) and a COX2 inhibitor (Etodolac), in order to attenuate the surgically induced immunosuppression and other physiological perturbations, aiming to reduce the rate of tumor recurrence and distant metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for surgery for primary resection of colon and rectal cancer in curative intent.
* Single colonic or rectal carcinoma, proofed by full colonoscopy and tumor biopsy. If colonoscopy failed to reach the cecum, proximal colonic investigation will be made using contract enema or CT colonography.
* No evidence of metastatic disease prior to surgery. Minimal workup would include abdominal CT with IV contrast (or CT+liver US) and chest XR.
* Age between 18 and 75 year old.
* ASA score of 1-3
* The patient is able to understand the study objectives and procedures, able to comply with the protocol, and is capable to sign an informed consent.

Exclusion Criteria:

* Patients with metastatic disease, known prior to surgery.
* Patients in whom metastatic disease is found at surgery will complete the intervention phase, followed for additional month for potential complications, and will exit the study to allow potential participation in further clinical trials.
* Patients in whom surgical resection is planned without curative intent.
* Patients with renal failure, measured by Creatinine level >1.5
* Patients with significant heart failure (NYH 3 or higher)
* Patients with significant liver failure (known cirrhosis, Bilirubin level>2)
* Patients suffering from asthma
* Patients with known allergy to one or more of the study medications
* Patients with known allergy to any medication from the non-steroidal anti-inflammatory drug group.
* Patients with diabetes (type 1 or 2).
* Patients treated chronically with one or more of the study medications
* Patients treated chronically with any type of Beta adrenergic blocker.
* Patients treated chronically with any type of COX inhibitor.
* Patients with second or third degree AV block.
* Patients with sinus bradycardia (patients with heart rate of less than 50).
* Patients with sick sinus syndrome.
* Patients with Prinzmetal's angina
* Patients with right sided heart failure owing to pulmonary hypertension.
* Patients with significant cardiomegaly
* Patients with (current) pheochromocytoma
* Patients with chronic Digoxin treatment
* Patients with active peptic disease
* Patients with peripheral vascular disease
* Patients with history or concomitant malignant disease of any type.
* Patients who were treated with chemotherapy in the last 10 years for any reason besides neo-adjuvant therapy for rectal cancer within the last six months.
* Pregnant woman.
* Patients participating in any other clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Rate of recurrent and metastatic cancer | 3 years

SECONDARY OUTCOMES:
magnitude and duration of surgically induced immune depression, as reflected in the blood samples | early postoperative
Early postoperative morbidity and mortality | 30 days

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Rabin- Beilinson Medical Center, Petah Tikva
  - Tel Aviv-Sourasky Medical Center, Tal Aviv
  - Sheba Medical Center, Tel Litwinsky

REFERENCES:
- [Derived] Hicks BM, Murray LJ, Powe DG, Hughes CM, Cardwell CR. beta-Blocker usage and colorectal cancer mortality: a nested case-control study in the UK Clinical Practice Research Datalink cohort. Ann Oncol. 2013 Dec;24(12):3100-6. doi: 10.1093/annonc/mdt381. Epub 2013 Sep 19. PMID 24050955